CLINICAL TRIAL: NCT04417608
Title: Looking for Minimum Dose to Induce Sympathectomy in Infraclavicular Brachial Plexus Block
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, anchihhsu, Principal Investigator, Taipei Medical University WanFang Hospital
Other Study IDs: N202003147
Record Dates: First submitted 2020-05-31; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Finding the Minimum Dose to Induce Sympathectomy in Infraclavicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Infraclavicular brachial plexus block — Ultrasound-guided infraclavicular brachial plexus block

SUMMARY:
For patients who undergoing hemodialysis, it is important to have good AV fistula. One third of AV fistula usually fail during early stage. It is helpful to use nerve block to dilate the blood vessels and enhance the prognosis. But 0.2% Ropivacaine usually cause muscle weakness in present studies. The investigators hope to find the lowest concentration to provide sympathectomy without muscle weakness. Because the patients with hemodialysis usually have multiple co-morbidity, thus we choose patients with forearm fracture at the first place. With this result, the investigators can design further study for patients with hemodialysis. The investigators prefer proximal approach because brachial plexus run together in the cosctoclavicular space and show lower incidence of incomplete work.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-80 y/o, BW: 40-90 kilograms，ASA class I-III，No pre-existing neuropathy，Scheduled for upper limb surgery.

Exclusion Criteria:

1. Pre-existing neuropathy (ex: polyneuropathy)
2. History of allergy to xylocaine、ropivacaine、epinephrine
3. Emergent surgery
4. Coagulopathy
5. Patient who can not express themselves

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled for upper limb surgery
Sampling Method: Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2020-06-04 (Estimated); Primary Completion 2021-07-04 (Estimated); Study Completion 2021-07-04 (Estimated)

PRIMARY OUTCOMES:
Change of diameter of basilic vein and brachial artery | Change from baseline diameter(pre-nerve block) at 45min
  Use ultrasound to measure the difference of diameter at different time point.
Change of diameter of basilic vein and brachial artery | Change from baseline diameter(pre-nerve block) at 24hour
  Use ultrasound to measure the difference of diameter at different time point.
Change of diameter of basilic vein and brachial artery | Change from baseline diameter(pre-nerve block) at 48hour
  Use ultrasound to measure the difference of diameter at different time point.

SECONDARY OUTCOMES:
Sensory block of upper limb | 45min post nerve block
  A validated 3-point scale was used: 0 = no block (patient has normal sensation), 1 = patient can feel cold, but the sensation is reduced compared with the unblocked side, and 2 = complete anesthesia.
Sensory block of upper limb | 24hour post nerve block
  A validated 3-point scale was used: 0 = no block (patient has normal sensation), 1 = patient can feel cold, but the sensation is reduced compared with the unblocked side, and 2 = complete anesthesia.
Motor block of upper limb | 45min post nerve block
  A validated 3-point scale was used: 0 = no block (patient has normal power), 1 = patient can feel weakness with the unblocked side, and 2 = complete anesthesia.
Motor block of upper limb | 24hour post nerve block
  A validated 3-point scale was used: 0 = no block (patient has normal power), 1 = patient can feel weakness with the unblocked side, and 2 = complete anesthesia.
Motor block of upper limb | 48hour post nerve block
  A validated 3-point scale was used: 0 = no block (patient has normal power), 1 = patient can feel weakness with the unblocked side, and 2 = complete anesthesia.